CLINICAL TRIAL: NCT06068192
Title: A Study on the Registration of Sepsis Patients in the Emergency Department of the First Hospital of Jilin University
Brief Title: Registration of Sepsis Patients in the Emergency Department
Acronym: RSP
Status: Not yet recruiting | Type: Observational
Sponsor: The First Hospital of Jilin University (Other)
Responsible Party: Sponsor
Other Study IDs: RSP
Record Dates: First submitted 2023-09-28; First posted 2023-10-05 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-09

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood,urine and other infection sites to detect the pathogen.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 28th day death group: Patient dies within 28 days after hospitalization
  Interventions: Other: no intervention
- non-28th day death group: The patient does not die within 28 days after hospitalization
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
1) Establish a clinical data database for sepsis patients in the Emergency Department of the First Hospital of Jilin University. Describe the clinical data and prognosis of patients with simple systemic inflammatory response syndrome (common infection), pre sepsis, sepsis, and septic shock. 2) Explore the risk factors related to the progression of sepsis in patients in the early stages, as well as the risk factors related to the patient's prognosis. 3) Analyze the risk factors related to the prognosis of sepsis patients, and provide clinical basis for the treatment and long-term prognosis of sepsis patients. 4) Search for diagnostic biomarkers and prognostic serum biomarkers for patients with sepsis, sepsis, and septic shock.

DETAILED DESCRIPTION:
The study site and population included patients with systemic inflammatory response syndrome caused by "infectious factors" who were admitted to the Emergency Department of the First Hospital of Jilin University from January 1, 2023 to December 31, 2027. The screening criteria for the study population were patients with "systemic inflammatory response syndrome" caused by sensory factors who were continuously registered and treated at the Emergency Department of the First Affiliated Hospital of Jilin University from January 1, 2023 to December 31, 2027. A. Inclusion criteria: 1) Age greater than or equal to 15 years old; 2) A patient who sought medical treatment at the Emergency Department of Jilin University First Hospital due to "systemic inflammatory response syndrome" (see relevant concepts and definitions in section 4.2 below). 3) Within 24 hours of seeking medical attention, evidence of "infection" can be clearly detected through imaging and laboratory examinations. Patients can be diagnosed and classified as at least one of the following conditions: respiratory system infection, digestive system infection, urinary system infection, blood borne infection, or skin soft tissue infection. B. Exclusion criteria: Patients with any of the following conditions need to be excluded from this study, including: 1) pregnant and lactating women; 2) Active pulmonary tuberculosis; 3) Patients who do not agree to participate in this study. The follow-up strategy is to follow up for 1 month and 3 months after discharge. Obtain patient information through telephone follow-up or on-site follow-up, with a loss of follow-up rate not exceeding 20%. The telephone follow-up includes the patient's daily discomfort symptoms, whether the infection has recurred, whether infection related symptoms have reappeared, if there is any organ damage upon discharge, it is necessary to inquire about re examination and recovery status, whether there are new diseases and treatment measures, and medication status; The follow-up at the hospital includes the patient's basic vital signs, blood routine, liver function, kidney function, cardiac ultrasound, and quality of life assessment. Please refer to the attachment for details< Table 3. Patient Follow up Information Collection Table>Follow up Time Range Follow up Method: 1 month before discharge, 1 week phone follow-up and/or hospital visit. 2 months after discharge, 1 week phone follow-up and/or hospital visit. Related concepts and definitions: A. Systemic Inflammatory Response Syndrome (SIRS) (refer to the 8th edition of Internal Medicine and the 2nd edition of Emergency Medicine), with the presence of corresponding injury factors, SIRS can be diagnosed if two or more of the following occur. 1) Body temperature>38 ℃ or<36 ℃. 2) Heart rate>90 beats per minute or hypotension (systolic blood pressure<90 mmHg, or a decrease of>40 mmHg from baseline). 3) Shortness of breath (>20 breaths/minute) or hyperventilation (PaCO2<32mmHg). 4) Peripheral blood white blood cell count greater than 12 × 109/L or less than 4 × 109/L, or immature white blood cells greater than 10%, but other reasons that can cause the aforementioned acute abnormal changes should be ruled out. B. Grouping of SIRS patients: The diagnostic criteria in this section refer to the 2021 Surviving sepsis campaign guidelines

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than or equal to 15 years old; 2) A patient who sought medical treatment at the Emergency Department of Jilin University First Hospital due to "systemic inflammatory response syndrome" (see relevant concepts and definitions in section 4.2 below). 3) Within 24 hours of seeking medical attention, evidence of "infection" can be clearly detected through imaging and laboratory examinations. Patients can be diagnosed and classified as at least one of the following conditions: respiratory system infection, digestive system infection, urinary system infection, blood borne infection, or skin soft tissue infection.

Exclusion Criteria:

1. pregnant and lactating women; 2) Active pulmonary tuberculosis; 3) Patients who do not agree to participate in this study.

Min Age: 15 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The study site and population included patients with systemic inflammatory response syndrome caused by "infectious factors" who were admitted to the Emergency Department of the First Hospital of Jilin University from January 1, 2023 to December 31, 2027. The screening criteria for the study population were patients with "systemic inflammatory response syndrome" caused by sensory factors who were continuously registered and treated at the Emergency Department of the First Affiliated Hospital of Jilin University from January 1, 2023 to December 31, 2027.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
The patient dies within 28 days after hospitalization | within 28 days after hospitalization
  The patient dies within 28 days after hospitalization
The patient does not die within 28 days after hospitalization | within 28 days after hospitalization
  The patient does not die within 28 days after hospitalization

IPD SHARING:
Plan to Share IPD: Undecided